CLINICAL TRIAL: NCT05717244
Title: Comparison of Two Pupillometer for Determining Pupil Diameter in Healthy Participants
Brief Title: Comparison of Two Different Pupillometer
Status: Completed | Type: Observational
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2WIN2023
Record Dates: First submitted 2023-01-29; First posted 2023-02-08 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2023-02

CONDITIONS: Measurement of Pupil Diameter
Keywords: 2WIN-S; scotopic pupil size

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: 2WIN-S — Determining pupil diameter by 2WIN-S
Device: OPD — Determining pupil diameter by OPD

SUMMARY:
With the development of refractive surgery, the size of scotopic pupil has been widely concerned by clinicians. Historically, the measurement of pupil size included the use of a pupil ruler, which is known for its drawback of being very subjective and lacking precision. While infrared pupillometry devices such as OPD-Scan III and Sirius are available for accurately and reliably measuring pupil size. Nevertheless, the aforementioned equipments are costly and cumbersome to move in terms of screening and field trial logistics settings. And 2WIN-S is a portable refractor, it can in a short period of diopter and scotopic pupil size and other data obtained at the same time. Therefore, the aim of this study was to compare the agreement between 2WIN-S and OPD-Scan III in measuring scotopic pupil size and the repeatability of 2WIN-S.

DETAILED DESCRIPTION:
Pupil diameter is a parameter of great interest in understanding brain systems and modern refractive surgery. Pupillometry, the measurement of variations in pupil dilation, has offered encouraging evidence for the involvement of disturbed reactivity in depression risk, according to studies. According to research, the pupil dilates in reaction to stimuli requiring a larger cognitive load or a greater emotional intensity. Importantly, studies have related pupil size variations to brain activity in regions associated with emotion regulation, including the dorsolateral prefrontal cortex (DPFC) and the agenesis of the corpus callosum (ACC) . Thus, pupillometry is proposed as a viable peripheral gauge for a variety of brain systems involved in the processing of emotional information.

Some of the postoperative complaints of patients having refractive corneal or lens surgery are related to visual quality and are associated with large pupils since optical aberrations become more dominant when the pupil dilates . If the pupil size exceeds the optical zone size, a marked increase in higher-order aberrations could be observed. Patients might complain about poor contrast sensitivity, increased glare disability, or halos. Precise measurement of scotopic pupil diameter has therefore become an essential step in the preoperative evaluation of patients suitable for refractive surgery and is an important inclusion or exclusion criterion.

This study aimed to assess the agreement and reproducibility of scotopic pupil size measurements using 2WIN-S compared with OPD-Scan III in Chinese adults.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* signed informed consent
* willing to participate in the study

Exclusion Criteria:

Exclusion criteria were ocular pathology known to interfere with pupillometer outcome and pupil abnormalities (eg: glaucoma, iritis, cataract, corneal scarring, any history of ocular surgery, and history of trauma.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adults attending ophthalmology clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Scotopic pupil size | 1 day
  Scotopic pupil size will be measured using 2WIN-S with OPD-Scan III.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel E Pazo, MD, PhD, Study Chair — He Eye Hospital, Shenyang, China
Locations (1):
- He Eye Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jones NP, Siegle GJ, Mandell D. Motivational and emotional influences on cognitive control in depression: A pupillometry study. Cogn Affect Behav Neurosci. 2015 Jun;15(2):263-75. doi: 10.3758/s13415-014-0323-6. PMID 25280561
- [Background] Siegle GJ, Steinhauer SR, Friedman ES, Thompson WS, Thase ME. Remission prognosis for cognitive therapy for recurrent depression using the pupil: utility and neural correlates. Biol Psychiatry. 2011 Apr 15;69(8):726-33. doi: 10.1016/j.biopsych.2010.12.041. PMID 21447417
- [Background] Siegle GJ, Granholm E, Ingram RE, Matt GE. Pupillary and reaction time measures of sustained processing of negative information in depression. Biol Psychiatry. 2001 Apr 1;49(7):624-36. doi: 10.1016/s0006-3223(00)01024-6. PMID 11297720
- [Background] Siegle GJ, Steinhauer SR, Stenger VA, Konecky R, Carter CS. Use of concurrent pupil dilation assessment to inform interpretation and analysis of fMRI data. Neuroimage. 2003 Sep;20(1):114-24. doi: 10.1016/s1053-8119(03)00298-2. PMID 14527574
- [Background] Critchley HD, Tang J, Glaser D, Butterworth B, Dolan RJ. Anterior cingulate activity during error and autonomic response. Neuroimage. 2005 Oct 1;27(4):885-95. doi: 10.1016/j.neuroimage.2005.05.047. PMID 15996878
- [Background] Urry HL, van Reekum CM, Johnstone T, Kalin NH, Thurow ME, Schaefer HS, Jackson CA, Frye CJ, Greischar LL, Alexander AL, Davidson RJ. Amygdala and ventromedial prefrontal cortex are inversely coupled during regulation of negative affect and predict the diurnal pattern of cortisol secretion among older adults. J Neurosci. 2006 Apr 19;26(16):4415-25. doi: 10.1523/JNEUROSCI.3215-05.2006. PMID 16624961
- [Background] Fardell J. Poverty and infant deaths. Nurs Times. 1989 Jan 11-17;85(2):18. No abstract available. PMID 2922323
- [Background] Martinez CE, Applegate RA, Klyce SD, McDonald MB, Medina JP, Howland HC. Effect of pupillary dilation on corneal optical aberrations after photorefractive keratectomy. Arch Ophthalmol. 1998 Aug;116(8):1053-62. doi: 10.1001/archopht.116.8.1053. PMID 9715686
- [Background] Rosen ES, Gore CL, Taylor D, Chitkara D, Howes F, Kowalewski E. Use of a digital infrared pupillometer to assess patient suitability for refractive surgery. J Cataract Refract Surg. 2002 Aug;28(8):1433-8. doi: 10.1016/s0886-3350(01)01350-5. PMID 12160815
- [Background] Liu Q, Yang X, Lin L, Liu M, Lin H, Liu F, Xie Y, Lam DSC. Review on Centration, Astigmatic Axis Alignment, Pupil Size and Optical Zone in SMILE. Asia Pac J Ophthalmol (Phila). 2019 Sep-Oct;8(5):385-390. doi: 10.1097/01.APO.0000580144.22353.46. PMID 31567265
- [Background] Couret D, Boumaza D, Grisotto C, Triglia T, Pellegrini L, Ocquidant P, Bruder NJ, Velly LJ. Reliability of standard pupillometry practice in neurocritical care: an observational, double-blinded study. Crit Care. 2016 Mar 13;20:99. doi: 10.1186/s13054-016-1239-z. PMID 27072310
- [Background] Nyholm B, Obling L, Hassager C, Grand J, Moller J, Othman M, Kondziella D, Kjaergaard J. Superior reproducibility and repeatability in automated quantitative pupillometry compared to standard manual assessment, and quantitative pupillary response parameters present high reliability in critically ill cardiac patients. PLoS One. 2022 Jul 28;17(7):e0272303. doi: 10.1371/journal.pone.0272303. eCollection 2022. PMID 35901103